CLINICAL TRIAL: NCT04664348
Title: Is the Positioning of the Lumbar Spine Relevant to the Manual Treatment of the Chronic Low Back Pain
Brief Title: Does Low Back Position Matters in Manual Therapy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2020/42
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Posteroanterior lumbar mobilization (extension of the lumbar spine) (Experimental)
  Interventions: Other: Posteroanterior mobilization (extension)
- Experimental: Posteroanterior lumbar mobilization (lumbar spine in neutral positioning) (Experimental)
  Interventions: Other: Posteroanterior mobilization (neutral)

INTERVENTIONS:
Other: Posteroanterior mobilization (neutral) — Positioning of the patient: Prone position with the lumbar area uncovered.
  Positioning of the therapist: Stand to one side of the table at the pelvis of the patient.
  Explanation of the technique: The contact will be made with the hypothenar eminence on the spinous processes to be treated. The other hand of the physiotherapist will reinforce the grip to obtain greater stability and precision. It will proceed to carry out some posteroanterior pushes of the target vertebrae, in order to desensitize the chosen area. The force exerted and the speed of the technique will be controlled by the therapist. The technique will be finished when the participant let the therapist know when the pain is gone or when the patient no longer refer a decrease on its pain.
  Both groups: The patient will be provided with a list of exercises focused on improving resistance to mechanical load in the lumbar region. The completion of the exercise will be in the 6 weeks of the duration of the treatment.
  Arms: Experimental: Posteroanterior lumbar mobilization (lumbar spine in neutral positioning)
Other: Posteroanterior mobilization (extension) — Positioning of the patient: Prone position with the lumbar area uncovered. The head of the stretcher will be raised upwards, placing progressively to extend the lumbar region, until the patient communicates the reproduction of its symptoms.
  Positioning of the therapist: Stand to one side of the table at the pelvis of the patient.
  Explanation of the technique: The contact will be made with the hypothenar eminence on the spinous processes to be treated. The other hand of the physiotherapist will reinforce the grip to obtain greater stability and precision. It will proceed to carry out some posteroanterior pushes of the target vertebrae, in order to desensitize the chosen area. The force exerted and the speed of the technique will be controlled by the therapist. The technique will be finished when the participant let the therapist know when the pain is gone or when the patient no longer refer a decrease on its pain.
  Arms: Experimental: Posteroanterior lumbar mobilization (extension of the lumbar spine)

SUMMARY:
The study will be carried out at the Faculty of Nursing and Physiotherapy of the University of Alcalá. The study has been approved by the Animal Research and Experimentation Ethics Committee of the University of Alcalá. A total of 46 subjects of legal age with non-specific chronic low back pain will be selected and randomized into two interventions.

The first group will receive lumbar posteroanterior mobilizations with the lumbar spine in extension and the second group will receive lumbar mobilizations with neutral position of the spine. Both groups will also receive a home exercise program for the lumbar spine.

The total duration of the treatments will be 6 weeks, with pre-treatment, at 3 weeks of the treatment, post-treatment evaluations at 6 weeks, with a follow-up after 1 month and with a follow-up after 3 months.

The objective will be to evaluate which of the two interventions is more effective in addressing disability variables (main variable), pressure pain threshold, pain location, pain intensity, quality of life, quality of sleep, depression and kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* subjects with unspecific low back pain of 3 or more months of evolution prior commencement of the intervention

Exclusion Criteria:

* lumbar pain related to infectious diseases
* fractures
* oncological processes
* women in gestation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in Disability | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  measured with the Oswestry Low Back Pain Disability Questionnaire. The interpretation of the scores of this scale varies from 0% to 100%.
  0% to 20%: minimal disability: The patient can cope with most living activities.
  21%-40%: moderate disability 41%-60%: severe disability 61%-80%: crippled 81%-100%: These patients are either bed-bound or exaggerating their symptoms.

SECONDARY OUTCOMES:
Changes in Pressure pain threshold | Baseline, 3 weeks and 6 weeks after intervention commencement
  measured with a Wagner brand Force Dial with a 1 cm2 rubber disc at the end of the device.
Changes in Site of pain | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  measured with the body pain map
Pain measured with visual analogic scale | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  A straight horizontal line of fixed length, usually 100 mm is drawn. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (worst) to the right (best).
Health measured with the short form health survey version II | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  It consists of 12 items from the 8 dimensions of the short form health survey 36: Physical Function, Function Social, Physical role, Emotional role, Mental health, Vitality, Body pain , General Health. For each of the 8 dimensions, the items are coded, aggregated and transformed into a scale that ranges from 0 (the worst state of health for that dimension) to 100 (the best state of health).
Quality of sleep measured with the Pittsburgh Sleep Quality Index | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  In scoring the Pittsburgh Sleep Quality Index, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Depression measured with Beck's Depression Inventory | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
  Higher total scores indicate more severe depressive symptoms.
Kinesiophobia measured with the TAMPA scale of kinesiophobia | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  The total score ranges between 17 and 68. A high value on the TAMPA scale of kinesiophobia indicates a high degree of kinesiophobia.
  Cutoff score developed by Vlaeyen:
  * score of 37 or over is considered as high
  * scores below 37 is considered as low)
Changes in Medication | Baseline, 3 weeks, 6 weeks, 1 month and 3 months after intervention commencement
  The patient will be asked about how many days a week they have needed to take medication

CONTACTS AND LOCATIONS:
Locations (1):
- Adrián Cabañas, Alcalá de Henares, Madrid, Spain